CLINICAL TRIAL: NCT01093274
Title: Efficacy and Safety of Polyethylene Glycol Compared With Sodium Picosulphate for Bowel Preparation Before Colonoscopy, a Prospective Randomized, Controlled Study
Brief Title: Efficacy and Safety of Polyethylene Glycol Compared With Sodium Picosulphate for Bowel Preparation Before Colonoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Eyal Gal MD, Rabin Medical Center- Beilinson hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Gal001
Record Dates: First submitted 2010-02-22; First posted 2010-03-25 (Estimated); Last update posted 2010-03-25 (Estimated); Status verified 2010-02

CONDITIONS: Bowel Preparation
Keywords: colonoscopy; Cathartics; Sodium picosulfate; Polyethylene Glycol
MeSH Terms: interventions — picosulfate sodium; Polyethylene Glycols

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Polyethylene glycol (Active Comparator): Preparation with Polyethylene Glycol and bisacodyl
  Interventions: Drug: Polyethylene Glycol
- Picolax (Experimental): Preparation with Sodium Picosulphate and Bisacodyl.
  Interventions: Drug: Sodium Picosulphate

INTERVENTIONS:
Drug: Sodium Picosulphate — 2 Sachets
  Arms: Picolax
Drug: Polyethylene Glycol — 3 Liters solution
  Other Names: Meroken new; Go-Lytely
  Arms: Polyethylene glycol

SUMMARY:
Patients intended for ambulatory colonoscopy will be randomized into 2 groups

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory patients scheduled for elective colonoscopy
* Age 18-80

Exclusion Criteria:

* Renal insufficiency (serum creatinine ≥2.0 mg/dl)
* Symptomatic congestive heart failure
* Recent myocardial infarction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients requiring repeat colonoscopy because of poor preparation | quality of preparation will be assessed during colonoscopy
  Quality of preparation: good, moderate, poor

SECONDARY OUTCOMES:
Patient's satisfaction as measured by questionnaire and willingness to repeat same preparation on future examination | Questionnaire will be filled before colonoscopy
  Patient satisfaction on questionnaire referring to taste, compliance with protocol, side effects, willingness to repeat preparation.

CONTACTS AND LOCATIONS:
Overall Officials: Eyal Gal, MD, Principal Investigator — Rabin Medical Center - Beilinson hospital
Locations (1):
- Rabin Medical Center - Beilinson Hospital, Petah Tikva, Israel